CLINICAL TRIAL: NCT00000117
Title: Intravenous Immunoglobulin Therapy in Optic Neuritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-13
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Immunoglobulins

INTERVENTIONS:
Drug: Immunoglobulin

SUMMARY:
To determine whether high-dose intravenous immunoglobulin (IVIg) is more effective than placebo in restoring lost visual function (visual acuity) in optic neuritis (ON).

To determine the time course of recovery following IVIg administration. If the reports of IVIg-associated clinical improvement occurring within 3 to 6 months following treatment can be confirmed, this would provide indirect evidence that IVIg may promote central nervous system (CNS) remyelination in optic neuritis and multiple sclerosis (MS).

DETAILED DESCRIPTION:
Optic neuritis is the leading cause of transient, spontaneous, reversible visual loss in young adults. Characteristically, patients present with central visual loss that peaks within a few days and is often associated with eye pain. Visual loss may be complete. Spontaneous recovery usually begins within 4 weeks, and marked recovery occurs within 1 to 3 months in most patients. Although clinical improvement is the rule, not all patients recover fully, and many are left with residual symptoms. Although there are limited pathological studies in inflammatory ON, the pathological changes are thought to be virtually identical with those seen in MS, with disruption of the blood-nerve (brain) barrier; primary demyelination with axonal sparing; variable degrees of lymphocytic infiltration; an abundance of macrophages around the inflammatory demyelination lesion; various degrees of remyelination; and, later, oligodendrocyte loss, axonal loss, and gliosis.

Remyelination by oligodendrocytes occurs early in the MS lesion, as documented by myelin sheaths that are abnormally thin relative to axon diameter. These thin myelin sheaths are often seen prominently at the edge of demyelinated plaques. A recent series of studies has shown that within weeks of the initial event, there is extensive oligodendrocyte regeneration and remyelination. These immature oligodendrocytes express a series of developmentally restricted antigens. This finding has been interpreted to suggest that the cells that repopulate the acute plaque and that affect remyelination are newly generated and not residual, mature oligodendrocytes. These observations support the possibility that factors that promote remyelination could be used to improve clinical recovery in ON and MS.

Work at the Mayo Clinic, has shown that both immunoglobulin G (IgG) directed against spinal cord antigens and purified polyclonal mouse IgG administered systemically promote extensive remyelination in SJL mice chronically infected with Theiler's virus. In addition, tissue culture studies suggest that IgG directed against CNS components may promote oligodendroglial proliferation and differentiation. Thus, experimental evidence exists for the concept that immunoglobulins may stimulate the proliferation and differentiation of oligodendrocytes. It is possible that myelin components on the surface of oligodendrocytes could function as receptors or components of receptors. Antibodies could mimic endogenous ligands, thereby inducing the proliferation or differentiation of these cells.

In a preliminary, open-label pilot study of patients with chronic, steroid-unresponsive ON, Drs. van Engelen, Hommes, and colleagues suggested that improvement in visual recovery could be seen following IgG treatment in patients with chronic, stable ON. These encouraging but preliminary basic and clinical studies have prompted us to design a double-blind and placebo-controlled clinical trial of IVIg in patients with recently acquired but apparently permanent muscle paralysis from MS (NS31506) and to develop this NEI-funded ON study (U10EY1096301).

In this randomized, placebo-controlled, double-blind clinical trial, 60 patients were assigned to receive either IVIg or a placebo over a period of 3 months. In order to be eligible, patients who meet the inclusion criteria needed to have a stable loss of visual function (unchanged between the pre-enrollment screening visit and the enrollment visit). All patients wre re-examined at 3, 6, 9, and 12 months, with the primary outcome being the impact of treatment on visual acuity at 6 months as determined by measurements on a retroilluminated Early Treatment Diabetic Retinopathy Study chart at 4 meters.

One group of patients received 0.4 g/kg Gammimmune N intravenously daily for 5 days, and thereafter once a month for 3 months (total: eight infusions). The other group of patients received infusions of 0.1 percent human serum albumin in 10 percent maltose (placebo) according to the identical protocol used for Gammimmune N.

The primary outcome measure was improvement in Logmar visual acuity by an average of 0.2 at 6 months. The secondary outcome measures included change in visual acuity at 3, 9, and 12 months, as determined on a retroilluminated ETDRS chart at 4 meters; change in visual fields at 6 and 12 months; change in visual evoked responses at 3, 6, and 12 months; and change in neurological examination (EDSS, FS, AI) at 3, 6, 9, and 12 months.

ELIGIBILITY:
To be eligible, patients must have a history of one or more episodes of previous demyelinating optic neuritis occurring in the setting of classic, adult-onset definite MS (clinically definite or laboratory-supported definite MS, or cranial MRI changes consistent with MS). In most cases, onset of MS will have occurred between the ages of 18 and 45. Patients must be younger than 50 years and must have apparently irreversible loss of visual acuity that meets the following criteria:

Visual acuity must be worse than 20/40 for at least 6 months. Patients must be able to read at least one letter on the 1-meter eye chart. Patients with no light perception or hand movement vision only are not eligible.

The above level of visual dysfunction must be observed on at least two serial examinations (separated by at least 1 month) in the Department of Ophthalmology at the Mayo Clinic.

Optic disc pallor must be present.

Patients must have impairment in the affected eye(s) on perimetry consistent with optic nerve dysfunction and must have a visual field mean deviation of less than -4.00.

Patients must not have received ACTH or corticosteroids within the preceding 2 months.

Max Age: 50 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 1995-08; Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Department of Neurology, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota